CLINICAL TRIAL: NCT00280748
Title: A Phase II Study of Treatment of Brain Metastases From Non-Small Cell Lung Cancer With Concurrent Whole Brain Radiation Therapy and Pemetrexed
Brief Title: Whole-Brain Radiation Therapy and Pemetrexed in Treating Patients With Brain Metastases From Non-Small Cell Lung Cancer
Acronym: NRR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0409; CDR0000551069 (Other: PDQ number)
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; tumors metastatic to brain
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study (Other): Single Arm Study
  Interventions: Drug: pemetrexed disodium; Radiation: radiation therapy

INTERVENTIONS:
Drug: pemetrexed disodium — 500 mg/m2 once every 21 days up to 126 days
  Other Names: Alimta
Radiation: radiation therapy — Patients will receive cranial irradiation at 2.5 Gy per fraction, 5 days a week, for 3 weeks to a total dose of 37.5 Gy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving radiation therapy together with pemetrexed may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving whole-brain radiation therapy together with pemetrexed works in treating patients with brain metastases from non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the response in patients with intracranial brain metastases from non-small cell lung cancer treated with whole-brain radiotherapy and pemetrexed disodium.

Secondary

* Determine the toxicity of this regimen in these patients.
* Estimate the overall survival of patients treated with this regimen.
* Evaluate the functional status of patients treated with this regimen.
* Assess neurological function and progression in patients treated with this regimen.
* Determine the response of patients with extracranial disease treated with pemetrexed disodium.

OUTLINE: Patients undergo whole-brain radiotherapy 5 days a week for 3 weeks beginning on day 1. Patients also receive pemetrexed disodium IV on day 1, 2, or 3 and day 28 of course 1, and on day 1 of each subsequent course. Treatment with pemetrexed disodium repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days and then every 2 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)
* Must have evidence of brain metastases by MRI or CT scan

PRIOR CONCURRENT THERAPY:

* Recovered from prior oncologic or major surgery
* Prior resection of all brain metastases or only site of brain metastases allowed provided there is radiologically evaluable intracranial metastases
* No prior cranial irradiation, including stereotactic radiosurgery
* More than 30 days since prior non-approved or investigational drug
* No other concurrent chemotherapy, immunotherapy, hormonal therapy, radiotherapy, surgery, or experimental medications

  * No single brain metastases or oligometastatic disease amenable to surgical resection or radiosurgery
* Relapsed NSCLC with brain metastases allowed
* Not a candidate for double-agent or platinum-based chemotherapy
* No leptomeningeal metastases
* No clinically relevant (defined by physical exam) pleural effusions or ascites that cannot be controlled with drainage or other procedures

Inclusion Criteria:

* Karnofsky performance status 70-100% OR ≥ 70 years of age
* Life expectancy > 3 months
* Absolute neutrophil count (ANC) > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin ≥ 8 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine clearance ≥ 45 mL/min
* Able to take vitamins, folic acid, and corticosteroids

Exclusion Criteria:

* Contraindication or intolerance to corticosteroid therapy
* Other malignancies within the past 5 years and disease-free OR prognosis is best defined by the NSCLC in the opinion of the attending physician
* Pregnant or nursing
* Positive pregnancy test
* Fertile patients must use effective contraception
* HIV positive
* Severe hypersensitivity to pemetrexed disodium
* Unable to discontinue NSAIDs for ≥ 5 days
* History of underlying dementia, Parkinson's disease, or Alzheimer's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Alamance Oncology/Hematology Associates, LLP, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00280748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 institutions between May 2005 and April 2008.
Period: Overall Study
Arm/Group | Single Arm Study
Started | 10
Completed | 6
Not Completed | 4
Not completed — Decline in performance | 3
Not completed — Extra-cranial disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 62.5 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Karnofsky Performance Status [Count of Participants; unit: Participants]
  KPS 90-100; minor symptoms of disease | 3
  KPS 80-90; some symptoms of disease | 0
  KPS 70-80; unable to carry on all normal activity | 6
  KPS unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Response of Intracranial Metastases (Complete and Partial Response)
Description: Radiographic response will be measured by RECIST, Response Evaluation Criteria In Solid Tumors Criteria, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 126 days
Population: Of the 10 patients, four patients were unevaluable due to extra-cranial disease progression or decline in performance status prevent re-evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 6
Participants
  partial response | 1
  stable disease | 3
  progressive disease | 2

2. Secondary Outcome: Number of Subjects Experiencing Adverse Events
Description: Toxicities was assessed using Common Terminology Criteria for Adverse Events (CTCAE) grading scale. Only toxicities with attribution to chemotherapy of "definite" or "probable" are considered, as determined by treating physician.
Time Frame: maximum 5 months
Population: All patients who received treatment were evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 10
Participants
  Anemia | 2
  Alpecia | 2
  Nausea | 6
  Anorexia | 1
  Pruritic rash on head | 1
  Cramps | 1
  Acute bronchitis | 1
  Blurred vision | 1
  Dry skin | 1
  Fatigue | 2

3. Secondary Outcome: Estimate the Overall Survival of Patients Treated With This Regimen.
Description: Patients were followed for survival from start of treatment until death from any cause (up to 4 years)
Time Frame: 4 years
Population: Four patients were unevaluable due to extra-cranial disease progression or decline in performance status preventing re-evaluation.
Measure: Median (Full Range); unit: months
Arm/Group | Single Arm Study
Number analyzed (Participants) | 6
months | 6.0 [1.7 to 8.3]

4. Secondary Outcome: Evaluate the Functional Status of Patients Treated With This Regimen.
Description: Functional status evaluated using the Karnofsky functional status scale. The Karnofsky Performance Scale (KPS) Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses. The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death.
Time Frame: baseline functional status only
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 10
Participants
  KPS 90-100; minor symptoms of disease | 3
  KPS 80-90; some symptoms of disease | 0
  KPS 70-80; unable to carry on all normal activity | 6
  KPS unknown | 1

5. Secondary Outcome: Neurological Function by Radiation Oncology Group (RTOG) Neurological Function Classification
Description: A classification score defined as follows:
  1. Able to work or to perform normal activities: neurological findings minor or absent
  2. Able to carry out normal activities with minimal difficulties. Neurological impairment does not require nursing care or hospitalization
  3. Seriously limited in performing normal activities. Requiring nursing care or hospitalization. Patients confined to bed or wheelchair or have significant intellectual impairment
  4. Unable to perform even minimal normal activities. Requiring hospitalization and constant nursing care and feeding. Patients unable to communicate or in coma.A higher score indicates worse function.
Time Frame: At Baseline, 30 days, and at end of treatment (maximum 5 months).
Population: This study was terminated due to slow enrollment and the planned statistical analyses could not be performed due to limit sample size. The data represents the results of patients enrolled and treated on the trial.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 10
scores on a scale
  Pre-Treatment | 1.6 [1 to 2]
  Cycle 2: number analyzed (Participants) | 9
  Cycle 2 | 1.9 [1 to 3]
  End of Treatment: number analyzed (Participants) | 6
  End of Treatment | 2.2 [1 to 3]

6. Secondary Outcome: Neurological Function by Mini Mental State Examination
Description: The Mini Mental State Examination is a 30-point questionnaire that is used to measure cognitive impairment. Score totals range from normal cognition (24-30 points), mild impairment (19-23 points), moderate impairment (10-18 points), to severe impairment (≤9 points).
Time Frame: Baseline (pre-treatment), 30 days (Cycle 2 Day 1), and maximum 5 months (end of treatment).
Population: This study was terminated due to slow enrollment and the planned statistical analyses could not be performed due to limited sample size. The data represents the results of patients enrolled and treated on the trial.
Measure: Mean (Full Range); unit: score on the scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 10
score on the scale
  Pre-Treatment | 28 [24 to 30]
  Cycle 2 Day 1 | 28.2 [25 to 30]
  End of treatment: number analyzed (Participants) | 6
  End of treatment | 27.7 [21 to 30]

7. Secondary Outcome: Response of Patients With Extracranial Disease Treated With Pemetrexed
Description: Response was measured by Response Evaluation Criteria In Solid Tumors RECIST criteria v1.0. Complete Response (CR) - Disappearance of all lesions Partial Response (PR) - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Stable Disease (SD) - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started. Progressive Disease (PD) - at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing nontarget lesions.
Time Frame: maximum 5 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 10
Participants
  partial response | 2
  stable disease | 3
  progressive disease | 1
  missing data | 4

ADVERSE EVENTS:
Time Frame: Adverse events were monitored up to 30 days after end of treatment
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 10/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=10)
pulmonary embolus (Vascular disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
hallucinations (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=10)
Right maxillary pain with drainage (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
face/upper/lower extremity swelling (Blood and lymphatic system disorders) | 1 (1)
swelling-lower extremities (Blood and lymphatic system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry Eyes (Eye disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Hemmorroids (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (1)
abdominal pain (General disorders) | 1 (1)
chest pain (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Hip pain (General disorders) | 1 (1)
left lower quadrant pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
rib cage pain (General disorders) | 1 (1)
right foot 4th toes numbness (General disorders) | 1 (1)
Acute bronchitis (Infections and infestations) | 1 (1)
UTI (Infections and infestations) | 1 (2)
difficulty sleeping (Metabolism and nutrition disorders) | 1 (1)
fatigue (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
weakness (Metabolism and nutrition disorders) | 2 (2)
weight loss (Metabolism and nutrition disorders) | 2 (2)
Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Nervous system disorders) | 2 (2)
Confusion (Nervous system disorders) | 3 (3)
depression (Nervous system disorders) | 2 (2)
Left eye visual disturbance (Nervous system disorders) | 1 (1)
memory impairment (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythemic/vesicular papule-right temple (Skin and subcutaneous tissue disorders) | 1 (1)
insect bite (Skin and subcutaneous tissue disorders) | 1 (1)
pruritic rash on head (Skin and subcutaneous tissue disorders) | 1 (1)
INR (Vascular disorders) | 1 (1)
Nosebleed (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes